CLINICAL TRIAL: NCT03442634
Title: Early Versus Traditional Oral Hydration After Cesarean Section; A Randomized Clinical Trial
Brief Title: Early Versus Traditional Oral Hydration After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Mohamed Mostafa, Obstetrics and Gynaecology Resident, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: cshydration
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Gastrointestinal Motility and Defecation Conditions
Keywords: bowel movements; cesarean section; oral hydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Hydration Group (Experimental): this study group will get 200 ml of sugar free water within 1 hour after cesarean section followed by oral hydration as per patients' desire then starting semisolid and solid foods when patients are open bowel Intervention: Early Oral Hydration
  Interventions: Other: Early Hydration
- Traditional Hydration Group (Active Comparator): this study group will get 200 ml of sugar free water after 6 hours after cesarean section followed by oral hydration as per patients' desire then starting semisolid and solid foods when patients are open bowel Intervention: Traditional Oral Hydration
  Interventions: Other: Traditional Oral Hydration

INTERVENTIONS:
Other: Early Hydration — this group will start oral hydration within 1 hour after cesarean section
  Other Names: Early Oral Hydration
  Arms: Early Hydration Group
Other: Traditional Oral Hydration — this group will start oral hydration 6 hours after cesarean section
  Other Names: Delayed Oral Hydration
  Arms: Traditional Hydration Group

SUMMARY:
this study helps us to compare and evaluate prospectively the benefits and safety of early hydration on bowel movement after cesarean section it includes two groups, a control group and a study group. the study group will get 200 ml of sugar free water within 1 hour after cs while the control group will get 200 ml of sugar free water 6 hours after cs

DETAILED DESCRIPTION:
Traditionally, patients are not given fluids or food after cesarean sections until bowel function returns as evidenced by bowel sounds, passage of stool or flatus since , uneventful (uncomplicated) cesarean sections have no effect on intestinal functions and with putting in minds the need of the mother for early hydration , movement , breast feeding and early discharge; that is why we are investigating the effectiveness and safety of early oral hydration after cesarean sections

ELIGIBILITY:
Inclusion Criteria:

* Term Singleton Pregnancy.
* Uncomplicated Elective Cesarean Section.
* Time of Cesarean Section doesn't exceed 90 minutes.
* Average blood loss during and after cesarean section (doesn't exceed 1000cc).
* All patients will be under spinal anesthesia.

Exclusion Criteria:

* Postpartum Hemorrhage.
* Surgical Complications Such as intestinal injury.
* Medical disorders such as Diabetes and Hypertension
* Factors that may influence postpartum blood loss as anemia, multiple pregnancy and polyhydraminos.
* Use of tocolytic drugs

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
audible intestinal sounds | first 12 hours after cesarean section
  auscultation of intestinal sounds hourly for the first 12 hours after cesarean section

SECONDARY OUTCOMES:
postoperative anorexia, nausea and vomiting | first 24 hours after cesarean section
  recording the incidence of git upset symptoms in the first 24 hours after cesarean section
time for first breast feeding | first 24 hours after cesarean section
  recording the time of first breast-feed
abdominal distension | first 24 hours after cesarean section
  recording the incidence of abdominal distension after cesarean section
amount of given intravenous fluids | up to 24 hours after cesarean section
  recording amount in ml of given iv fluids
need for pain analgesics | up to 24 hours after cesarean section
  recording the amount of pain analgesia needed after cesarean section
length of hospital stay | up to 48 hours after cesarean section
  recording the length of patients' stay at hospital
satisfaction measured with a visual analogue scale before patient discharge | first 6 hours after cesarean section
  measuring satisfaction level after cesarean section
time to first flatus | up to 48 hours after cesarean section
  recording the time at which the patient had its first flatus
time to first bowel movement | up to 72 hours after cesarean section
  recording the time at which the patient had her first bowel motion

CONTACTS AND LOCATIONS:
Overall Officials: Bassem A Islam, Lecturer, Study Director — Ain Shams Maternity Hospital; Karim A Wahba, Professor, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No